CLINICAL TRIAL: NCT06755086
Title: TF-antigen Targeting Molecular Probe for PET Imaging in Solid Tumors
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2024YJZ123
Record Dates: First submitted 2024-12-24; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Solid Tumors
Keywords: Solid Tumors; TF-antigen; CD176; PET imaging
MeSH Terms: interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 124I-hJAA-F11: All enrolled participants will be allocated to this arm (single-arm study). Study participants will undergo 124I-hJAA-F11 PET/CT scan.
  Interventions: Drug: 18-FDG

INTERVENTIONS:
Drug: 18-FDG — All study participants will undergo one 18F-FDG PET/ CT scan.

SUMMARY:
The objective of the study is to construct a noninvasive approach using 124I-labeled monoclonal antibody radiotracer to detect the Thomsen-Friedenreich antigen (TF-antigen, CD176) expression of tumor lesions in patients with solid tumors and to identify patients benefiting from TF-antigen targeting treatment.

DETAILED DESCRIPTION:
Analysis plan: 1. Recruit 3-5 participants to analyze preliminary pharmacokinetic/first-in-human dose (FIH), major organ distribution, and tumor uptake information via whole-body PET/CT imaging; 2. Recruit 20 participants to analyze in vivo safety and tumor targeting information; 3. Recruit all participants for a final summary.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 75 years, male or female;
2. ECOG performance status score of 0 or 1;
3. Expected survival time ≥ 6 months;
4. At least one measurable tumor lesion exists according to RECIST 1.1 criteria (e.g., lung cancer, gastric cancer, colorectal cancer, breast cancer, pancreatic cancer, hepatocellular carcinoma). The lesion must be eligible for biopsy within one month before or after a PET scan, and the patient must be able to provide 2-3 tissue slices of the lesion;
5. Subjects must fully understand and voluntarily agree to participate in the study and sign an informed consent form.

Exclusion Criteria:

1. Pregnant or breastfeeding women, or women planning to become pregnant during the study period or within three months after drug administration, as well as individuals donating sperm or eggs;
2. Individuals known or suspected to be allergic to the investigational drug or any of its components;
3. Individuals with significantly impaired liver or kidney function;
4. Individuals unable to comply with PET examinations or those with conditions such as claustrophobia that prevent them from undergoing PET scans.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Malignant tumor patients or suspected patients
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-01-06 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value（SUV） | 2 years
  SUV is a semi-quantitative analysis index to describe the radioactive uptake of lesions, which has certain reference value for differentiating benign and malignant lesions. The uptake of the tracer （124I-hJAA-F11） in solid tumor lesions by measuring SUV on PET/CT.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No